CLINICAL TRIAL: NCT01737515
Title: Investigation of Waist Circumference and Waist/Hip Ratio as a Predictive Risk Factor for Morbidity and Mortality After Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: AbdoWaistHip
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Main group: Consecutive patients undergoing colorectal surgery for benign or malignant colorectal disease without any diversion from the standard of care
  Interventions: Other: Abdominal waist and hip circumference

INTERVENTIONS:
Other: Abdominal waist and hip circumference — Abdominal waist and hip circumferences are measured clinically with a ruler as part of the standard pre-operative physical examination

SUMMARY:
Despite advances in surgical technique, preoperative patient evaluation and post-operative care, elective colorectal surgery carries a risk of mortality of approximately 2% and a morbidity rate ranging from 20-40%. Risk prediction is important for two reasons: it informs decision-making in individual cases before surgery (part of informed consent) and allows the comparison of actual outcome with predicted outcome. A number of scoring systems for assessing risk of death after surgery have been developed. They vary from simple scores based on a few variables to highly complex mathematical models requiring detailed data input. Recently, the Association Française de Chirurgie conducted a multicentre study to develop and validate a 4-item predictive score of mortality after colorectal resection which has good predictive value and is simple to use.

Although many surgeons associate obesity with adverse outcomes, recent large, well-designed studies have been unable to show that obesity (defined as Body Mass Index (BMI) >30) is an independent risk factor for major morbidity or mortality after general abdominal surgery. Recently abdominal obesity (waist measurement >102cm in men and >88cm in women) has been shown to have better correlation with cardiovascular disease than BMI and is strongly associated with a clustering of risk factors for cardiovascular disease and diabetes (insulin resistance, hyperglycaemia, hypertension, dyslipidaemia and abdominal obesity) known as the metabolic syndrome. Waist circumference and waist/hip ratio are measures of abdominal obesity that correlate with the amount of intra-abdominal rather than subcutaneous or general body fat and may be a better measure of the risk of intra-operative complications and post-operative morbidity following abdominal surgery than BMI.

The study will be prospective and multicentred, with 28 participating units in Belgium, France, Switzerland and Sweden. The coordinating centre will be UCL St Luc. The study will start on 1st September 2008 and will aim to include a minimum of 1000 patients. Consecutive patients undergoing elective colorectal resectional surgery for cancer or diverticulitis will be included. In addition to normal preoperative assessment, waist and hip circumference will be measured before surgery and specific data will be collected on intra and post-operative complications and mortality. Data will be recorded using an encrypted, anonymous database using variables carefully selected to assess short and long term outcomes. The study will be the first of its kind to investigate abdominal obesity as a predictive risk factor for colorectal surgery and will also be one of the biggest prospective studies of morbidity after colorectal surgery.

The aims of the study are a) to assess if waist measurement or waist/hip ratio is a better predictive risk factor for complications or mortality after colorectal surgery than BMI, and b) if this measurement adds accuracy to the AFC score in risk prediction.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer
* diverticulitis
* colonic volvulus
* colorectal polyp

Exclusion Criteria:

* Age < 18 years
* Inability to give informed consent
* Emergency surgery
* Pregnancy
* Comorbidity resulting in altered abdominal circumference measurement:

ascites secondary to chronic liver disease peritoneal carcinomatosis intestinal obstruction abdominal mass lesions >20cm diameter on CT scan. pre-existing abdominal stoma incisional hernia

* Inflammatory bowel disease: it is recognised that this group of patients carries a well-recognised increased risk of a number of adverse outcomes (e.g. venous thrombo-embolism) and elevated inflammatory parameters therefore it is proposed to exclude this group from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for whom elective colorectal resectional surgery (open and laparoscopic) is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 1415 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Morbidity after colorectal surgery | 30 days postoperatively
Mortality after colorectal surgery | 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Alex H Kartheuser, MD, PhD, MSc, Study Chair — Colorectal Surgery Unit, Cliniques universitaires Saint-Luc